CLINICAL TRIAL: NCT06151574
Title: Beamion LUNG 2: A Phase III, Open-label, Randomized, Active-controlled, Multi-centre Trial Evaluating Orally Administered Zongertinib (BI 1810631) Compared With Standard of Care as First-line Treatment in Patients With Unresectable, Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Harbouring HER2 Tyrosine Kinase Domain Mutations
Brief Title: Beamion LUNG-2: A Study to Test Whether Zongertinib (BI 1810631) Helps People With Advanced Non-small Cell Lung Cancer With HER2 Mutations Compared With Standard Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0008; 2023-504308-27-00 (Registry Identifier: CTIS); U1111-1294-1407 (Other: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer, Non-squamous, Non-small Cell
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental treatment arm (Experimental): zongertinib only
  Interventions: Drug: zongertinib
- Comparator arm (Active Comparator): pembrolizumab plus platinum-pemetrexed chemotherapy
  Interventions: Drug: pembrolizumab; Drug: cisplatin; Drug: carboplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: zongertinib — zongertinib
  Other Names: BI 1810631, Hernexeos®
  Arms: Experimental treatment arm
Drug: pembrolizumab — pembrolizumab
  Other Names: Keytruda®
  Arms: Comparator arm
Drug: cisplatin — platinum-pemetrexed chemotherapy
  Arms: Comparator arm
Drug: carboplatin — platinum-pemetrexed chemotherapy
  Arms: Comparator arm
Drug: pemetrexed — platinum-pemetrexed chemotherapy
  Arms: Comparator arm

SUMMARY:
This study is open to adults 18 years and older with advanced or metastatic non-small cell lung cancer. People can join the study if they have tumours with HER2 mutations and have not yet received any systemic therapy including chemotherapy for advanced or metastatic lung cancer. The purpose of this study is to find out whether a medicine called zongertinib (BI 1810631) can slow down the worsening of advanced non-small cell lung cancer better than the standard treatment available. Zongertinib may slow cancer cell growth by inhibiting HER2. This would prolong cancer re-occurrence and increase survival. Current standard treatment is pembrolizumab plus platinum-pemetrexed chemotherapy.

Participants are put into 2 groups by chance. One group receives zongertinib at regular times throughout the study and the other group receives infusions of pembrolizumab, pemetrexed and cisplatin or carboplatin (pembrolizumab plus platinum-pemetrexed chemotherapy) into a vein.

Participants may be in the study up to a maximum of 70 months. During this time, they visit the study site about every 3 weeks for study procedures. The doctors regularly check the size of the tumour with a CT or MRI scan, at the beginning of the study and every 6 weeks. After 18 months they check the tumour size every 12 weeks. Doctors regularly check whether the cancer has spread to other parts of the body. The doctors also regularly check participants' health and take note of any unwanted effects. The time it takes for the cancer to worsen is compared between the 2 groups to see whether the treatment works. The participants also fill in questionnaires about their symptoms and quality of life.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent form (ICF) in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
2. Patients ≥18 years of age or over the legal age of consent in countries where that is greater than 18 years at the time of signature of the ICF.
3. Histologically or cytologically confirmed diagnosis of an advanced and/or metastatic non-squamous Non-small cell lung cancer (NSCLC).
4. Documented Human epidermal growth factor receptor 2 (HER2) mutation in the Tyrosine kinase domain (TKD) as per local lab results.
5. An archival tumor tissue sample must be submitted to the central laboratory after inclusion of the patient to retrospectively confirm the HER2 status. If no archival tissue is available, this may be acceptable in exceptional cases after written agreement with the sponsor.
6. Patients who have not received any systemic treatment for unresectable, locally advanced or metastatic disease and are not eligible for curative therapy.
7. Presence of at least one measurable lesion according to Response evaluation criteria in solid tumors (RECIST) 1.1, as determined by the local site investigator/radiology assessment.
8. Eligible to receive treatment with the selected platinum-based doublet-chemotherapy (i.e. cisplatin/pemetrexed or carboplatin/pemetrexed) and pembrolizumab in accordance with the Summaries of Product Characteristics (SmPC)/Product Information.

Further inclusion criteria apply.

Exclusion criteria:

1. Previous or concomitant malignancies other than the one treated in this trial within the last 5 years, except;

   * effectively treated non-melanoma skin cancers
   * effectively treated carcinoma in situ of the cervix
   * effectively treated ductal carcinoma in situ
   * other effectively treated malignancy that is considered cured by local treatment
2. Tumors with targetable alterations with approved available therapy.
3. Lung-specific intercurrent clinically significant severe illness based on investigators assessment.
4. Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
5. Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to randomization or planned within 6 months after screening, e.g. hip replacement.
6. Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the trial or interfere with the evaluation of the safety and efficacy of the test drug.
7. History or presence of cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of ≥ III or IV, unstable angina or poorly controlled arrhythmia which are considered as clinically relevant by the investigator. Myocardial infarction, stroke, or pulmonary embolism within 6 months prior to randomization.
8. Any clinically important abnormalities (as assessed by the investigator) in rhythm, conduction, or morphology of resting electrocardiograms, e.g. complete left bundle branch block, third degree heart block.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-01-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 determined by blinded central independent review | up to 4 years and 5 months
  PFS is defined as the time from randomization until tumor progression according to RECIST 1.1 or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Key secondary endpoint: Overall Response (OR) according to RECIST 1.1 determined by blinded central independent review | up to 53 months
  OR is defined as confirmed best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to RECIST 1.1 from date of randomization until the earliest of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up or withdrawal of consent.
Key secondary endpoint: Change from baseline to Week 25 of Non-small cell lung cancer Symptom Assessment Questionnaire (NSCLC-SAQ) total score | at baseline, at week 25
  The NSCLC-SAQ is a 7-item patient-reported outcome measure for use in adults to assess symptoms of advanced NSCLC.
  It contains five domains and accompanying items that were identified as symptoms of NSCLC: cough (1 item), pain (2), dyspnea (1), fatigue (2), and appetite (1).
  The (total) lowest score possible is 0, and the highest (total) score possible is 20. Higher scores indicate more severe symptoms.
Key secondary endpoint: Overall Survival (OS) | up to 53 months
  OS is defined as the time from randomization until death from any cause.
Duration of response (DoR), determined by blinded central independent review | up to 53 months
  DoR is defined as the time from first documented complete response (CR) or partial response (PR) until the earliest of disease progression or death among patients with objective response.
PFS determined by blinded central independent review | up to 53 months
  PFS is defined as the time from randomization until tumor progression or death from any cause, whichever occurs earlier.
Bi-compartmental PFS, determined by blinded central independent review | up to 53 months
  Bi-compartmental PFS is defined as the time from randomization until tumor progression according to RECIST 1.1 or death from any cause, whichever occurs earlier.
OR determined by blinded central independent review | up to 53 months
  OR is defined as confirmed best overall response of CR or PR, from date of randomization until the earliest progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up or withdrawal of consent.
Change from baseline to Week 25 in the NSCLC-SAQ pain domain score | at baseline, at week 25
  The individual NSCLC-SAQ items use a five-point verbal rating scale from "No <symptom> At All" to "Very severe <symptom>" or from "Never to Always," corresponding to an (item) score of 0 to 4. A higher score indicates more severe symptoms.
Change from baseline to Week 25 in the NSCLC-SAQ dyspnea domain score | at baseline, at week 25
Change from baseline to Week 25 in the NSCLC-SAQ cough domain score | at baseline, at week 25
Change from baseline to Week 25 in the NSCLC-SAQ appetite domain score | at baseline, at week 25
Change from baseline to Week 25 in the NSCLC-SAQ fatigue domain score | at baseline, at week 25
Change from baseline to Week 25 in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) physical functioning domain score | at baseline, at week 25
  The EORTC QLQ-C30 is a quality of life questionnaire. It ranges from 0 to 100, higher scores equal worse outcome.
Occurrence of adverse events (AEs) during the on-treatment period, graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | up to 53 months
Occurrence of serious AEs (SAEs) during the on-treatment period, graded according to CTCAE version 5.0 | up to 53 months

CONTACTS AND LOCATIONS:
Locations (162):
- United States (22):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Pioneer Research Center - Bullhead City, Bullhead City, Arizona
  - Precision NextGen Oncology, Beverly Hills, California
  - ClinRé 001-022 (Premier Cancer Care and Infusion Center), Fresno, California
  - OPN Healthcare, Inc., Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - St. Louis Cancer Care, LLP, Bridgeton, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Cancer Care Specialists, Reno, Nevada
  - Northwell Health, Lake Success, New York
  - Montefiore Medical Center, The Bronx, New York
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Carolina Blood and Cancer Care Associates, PA, Rock Hill, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Cancer Institute, Edmonds, Washington
  - Swedish Cancer Institute, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
- Argentina (5):
  - Clinica Adventista Belgrano, CABA
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autónoma de Bs As
  - Instituto Oncologico de Cordoba, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
- Australia (5):
  - Prince of Wales Hospital-Randwick-66496, Randwick, New South Wales
  - Royal North Shore Hospital-St Leonards-20807, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Health, Heidelberg, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Austria (2):
  - Krems University Hospital, Krems
  - Clinic Floridsdorf, Vienna
- Belgium (3):
  - Brussels - HOSP Jules Bordet, Anderlecht
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (7):
  - Associacao Dr. Bartholomeu Tacchini, Bento Gonçalves
  - Hospital do Cancer de Londrina, Londrina
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - OncoClinicas Rio de Janeiro, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - ICESP - Instituto do Cancer do Estado de Sao Paulo, São Paulo
- Bradford Hill- Centro de Investigación Clínica, Recoleta, Chile
- China (16):
  - Cancer Hospital of Chinese Academy of Medical Science, Beijing
  - Beijing Cancer Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hospital, Zhengzhou
- France (9):
  - HOP Louis Pradel, Bron
  - CTR Leon Berard, Lyon
  - HOP Nord, Marseille
  - HOP Tenon, Paris
  - INS Curie, Paris
  - HOP Pontchaillou, Rennes
  - HOP Civil, Strasbourg
  - Hôpital Larrey - CHU de Toulouse, Toulouse
  - INS Gustave Roussy, Villejuif
- Germany (8):
  - Universitätsklinikum Augsburg, Augsburg
  - Gemeinschaftskrankenhaus Havelhöhe gGmbH, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Justus-Liebig Universität Gießen, Giessen
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Pius-Hospital, Oldenburg, Oldenburg
  - Universitätsklinikum Tübingen, Tübingen
- Hong Kong (3):
  - Queen Elizabeth Hospital-Hong Kong-51727, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Israel (4):
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Istituto Tumori Giovanni Paolo II, Bari
  - Istituto Di Candiolo, Candiolo (TO)
  - AOU Policlinico G. Rodolico San Marco, Catania
  - Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli
  - Azienda Ospedaliera Unversitaria di Parma, Parma
  - AOU Policlinico Umberto I, Roma
  - A. O. Ospedale Circolo Fond. Macchi, Varese
- Japan (20):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - Hirosaki University Hospital, Aomori, Hirosaki
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Shikoku Cancer Center, Ehime, Matsuyama
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hakodate Goryoukaku Hospital, Hokkaido, Hakodate
  - Hokkaido Cancer Center, Hokkaido, Sapporo
  - Kanazawa University Hospital, Ishikawa, Kanazawa
  - St. Marianna University Hospital, Kanagawa, Kawasaki
  - Kanagawa Cancer Center, Kanagawa, Yokohama
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Miyagi, Sendai
  - Okayama University Hospital, Okayama, Okayama
  - Osaka International Cancer Institute, Osaka, Osaka
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - Komagome Hospital, Tokyo, Bunkyo-ku
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Mexico (3):
  - Health Pharma Professional Research S.A. de C.V., Mexico City
  - Instituto Nacional de Cancerologia, México
  - FAICIC S de RL de C.V., Veracruz
- Netherlands (2):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek Amsterdam (METC AVL), Amsterdam
  - Maastricht University Medisch Centrum, Maastricht
- Norway (2):
  - Vestre Viken HF, Drammen Sykehus, Drammen
  - Oslo Universitetssykehus HF, Radiumhospitalet, Oslo
- Poland (4):
  - Polish Mother's Memorial Hospital - Research Institute, Lodz
  - Greater Poland Center of Pulmonology and Thoracic Surgery, Poznan
  - MED POLONIA SP Z O O, Clinical Trials Department,Poznan, Poznan
  - Oncology Center-Maria Sklodowska-Curie Institute, Warsaw
- Portugal (3):
  - Hospital CUF Tejo, Lisbon
  - Centro Hospitalar Lisboa Norte Hospital Pulido Valente, Lisbon
  - Hospital CUF Porto, Porto
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico
- Singapore (2):
  - National University Hospital-Singapore-22806, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (8):
  - Chungbuk National University Hospital, Cheongiu
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, St.Vincent's Hospital, Suwon
- Spain (13):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (5):
  - Western General Hospital, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - Guy's Hospital, London
  - The Royal Marsden Hospital, Chelsea, London
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency